CLINICAL TRIAL: NCT01798069
Title: Impact of an Educational Program 'Narrative Medicine (Workshop Reflexive Writing) ' Dedicated to Medical Students. A Randomized Controlled Trial.
Brief Title: Impact of Narrative Medicine (Workshop Reflexive Writing)
Acronym: INAMERE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RAV001
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2013-02

CONDITIONS: Empathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral intervention (Experimental): Students allocated to the experimental arm will follow 5 sessions in Class-led instruction of reflexive writing workshops. They will be divided into 12 sub-groups of 8 students. They will write their stories about their own experiences or the experiences of their family / patient.
  Interventions: Behavioral: reflective writing
- behavoral intervention (Active Comparator): Students allocated to the active comparator arm will follow 5 sessions in Class-led instruction of reading medical publication workshops. They will be divided into eight subgroups of 12 students. The first and fifth sessions will be presential, and 2nd 3rd and 4th sessions will be homework to do on internet.
  Interventions: Behavioral: reading medical publication workshops

INTERVENTIONS:
Behavioral: reflective writing — Students allocated to the experimental arm will follow 5 sessions in Class-led instruction of reflexive writing workshops. They will be divided into 12 sub-groups of 8 students. They will write their stories about their own experiences or the experiences of their family / patient.
  Arms: Behavioral intervention
Behavioral: reading medical publication workshops
  Arms: behavoral intervention

SUMMARY:
Objective: The aim of this study is to assess the impact of an educational program of Narrative Medicine "workshop reflexive writing "dedicated to medical students on the satisfaction of standardized patients.

Design: Randomized Controlled Trial in 2 arms. Participants: Medical students (4th years) of the University Paris Descartes. Methods: Participants will be randomized in two groups. The allocation of participants will be done by a computerized randomization list, the sequence will be created by an independent statistician. Participants will be blinded of the study hypothesis. Allocation concealment will be provided because only the statistician will have access to the randomization list.

A program of Narrative Medicine in Class-led instruction "workshop reflexive writing "vs "workshop reading medical publication".

Outcome: The primary endpoint will be the satisfaction of standardized patient relative to the empathy of the medical students. The secondary endpoints will be the empathy of the medical students; recommendation of the student by the standardized patients to friends or relatives; students' satisfaction.

Potential interests: The investigators believe that the workshop "reflexive writing" can develop the thinking of the student with respect to his behavior with the patient, and so the relation between student and patient.

ELIGIBILITY:
Inclusion Criteria:

* All students in the fourth year of medical school have chosen for their first 2 quarters to complete an internship in clinical hospital departments (i.e. where direct contact with patients)

Exclusion Criteria:

* All students refusing to participate in the study.
* All students repeaters.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
satisfaction of standardized patient will be assessed through the questionnaire recommended by the American Board of Internal Medicine (ABIM). | 5 months after randomization (i.e. 1 month after the end of the intervention)
  It consists of ten questions, denoted by EVGFP scale (excellent = 5, very good = 4, good = 3, fair = 2, poor = 1).

SECONDARY OUTCOMES:
The Jefferson Scale of Physician Empathy | 5 months after randomization (i.e. 1 month after the end of the intervention)
  self-administered questionnaire consisting of 20 items scored by a Likert-type scale (strongly agree = 7, strongly disagree = 1): 10 items are rated positively, others 10 items are rated negatively. The total score ranges from 20 to 140.

OTHER OUTCOMES:
The Interpersonal Reactivity Index | 5 months after randomization (i.e. 1 month after the end of the intervention)
  self-administered questionnaire with 4 subscales (Perspective Taking, Empathic Concern, Fantasy, Personal Distress) each containing seven items (a total of 28 items). The items are scored by a Likert scale (0 = Does not describe me well to 4 = Describes me very well).
students' satisfaction | 4 months after randomization (i.e. 1 month after the end of the intervention)
  measure on a numeric scale from 0 (without interest) to 10 (very interesting)
recommendation of the student by the standardized patient, to friends or relatives | 5 months after randomization (i.e. 1 month after the end of the intervention)
  : measure on a numeric scale from 0 (not at all) to 10 (entirely)

CONTACTS AND LOCATIONS:
Overall Officials: Francois GOUPY, Professeur, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Centre d'Epidémiologie Clinique, Assistance Publique, Hôtel Dieu, Paris, France